CLINICAL TRIAL: NCT04033120
Title: Making an Early Diagnosis of Talaromycosis - a Strategy to Reduce Morbidity and Mortality in Advanced HIV Disease in Southeast Asia
Brief Title: Making an Early Diagnosis of Talaromycosis Using a Novel Antigen Test
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Oxford University Clinical Research Unit, Vietnam (Other); National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102384
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: AIDS/HIV - RelatedDisease Associated With AIDS
Keywords: HIV; talaromycosis; endemic mycoses; opportunistic infections; penicilliosis; Southeast Asia
MeSH Terms: conditions — talaromycosis; Opportunistic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1: Symptomatic hospitalized patients: 900 patients admitted to the participating hospitals whom doctors suspect to have an infection and will perform TmAg testing alongside routine diagnostics and the following additional diagnostics:
  1. MycoF/lytic blood culture system
  2. Fujifilm lateral flow urine lipoarabinomannan (LF-LAM) test for tuberculosis
  3. Cryptotoccoal antigen in sera (CrAg) LFA for cryptococcosis
  4. Histoplasma antigen in urine (HAg) LFA for histoplasmosis
  We will follow patients closely for early diagnosis and treatment of culture confirmed talaromycosis over a six-month follow up period
- Cohort 2: Cohort 2: Asymptomatic outpatients: 500 patients registered at the outpatient clinics at the participating hospitals whom doctors do not suspect of having an active infection and will perform TmAg testing alongside the following diagnostics:
  1. CrAg LFA for cryptococcosis
  2. HAg LFA for histoplasmosis
  We will follow patients closely for early diagnosis and treatment of culture confirmed talaromycosis over a twelve-month follow up period.

SUMMARY:
This is a research study to determine whether a new antigen detection test called Mp1p EIA can make an early diagnosis of talaromycosis from the blood and urine of patients. Talaromycosis is a life-threatening infection caused by a fungus endemic in Southeast Asia commonly found in patients with advanced HIV disease called Talaromyces marneffei.

DETAILED DESCRIPTION:
This study aims to determine the diagnostic and prognostic values and the clinical impact of Talaromyces marneffei antigenemia (TmAg) in patients with advanced HIV disease using a novel enzyme immunoassay (EIA) detecting Tm-specific cell wall mannoprotein Mp1p. The data generated will be used to inform the design of future diagnostic clinical trials to test the utility of screening and providing pre-emptive antifungal therapy to prevent disease and reduce HIV mortality in Southeast Asia.

The primary objective is to screen for TmAg and determine its diagnostic and prognostic performance in symptomatic and asymptomatic HIV-infected patients with a CD4 count ≤100 cells/mm3.

We will test the following hypotheses:

1. In symptomatic hospitalized patient Cohort 1, the sensitivity of the Mp1p EIA will be higher than conventional culture method while simultaneously specificity is higher than 95% for diagnosing culture-confirmed talaromycosis over a six-month follow up period
2. In asymptomatic outpatient Cohort 2, there will be at least 30% difference in risk of talaromycosis development in TmAg-positive patients compared to TmAg-negative patients over a twelve-month follow up period
3. TmAg concentration predicts development of talaromycosis

Secondary Objectives include:

1. To assess the impact of presence of TmAg on clinical outcomes, including development of culture-confirmed talaromycosis, incidence of state III and IV AIDS events, subsequent hospitalizations, and death over six- to twelve-month follow up periods
2. To compare the diagnostic values of the Mp1p EIA when performed in plasma, sera, and urine samples and when performed in these matrices in combination

   We will test the following hypotheses:
3. To model the health economic benefits of screening and pre-emptive treatment for pre-clinical infection
4. To assess impact on clinic outcomes of screening all patients for cryptococcosis and histoplasmosis
5. To collect additional blood samples and store left-over samples for future research to validate infectious disease diagnostics and research to understand genetic susceptibility to infectious diseases relevant to HIV population

Participants in the study, will be asked questions about their medical and travel history. Participants will have blood and urine collected for the Mp1p EIA test to look for early talaromycosis infection and for other tests to look for common HIV-associated infections including tuberculosis, cryptococcosis, and histoplasmosis. They will be examined by a study doctor at least once weekly if they are in the hospital and will be followed in clinic monthly for between 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection (at least 2 of 3 HIV antibody tests are positive), AND
2. HIV-infected age ≥18 years, AND
3. CD4 count ≤100 cells/mm3 within the past 3 months, AND
4. Antiretroviral therapy (ART) naïve OR recent ART ≤3 months OR suspected or confirmed treatment failure on ART ≥12 months (defined as poor treatment adherence, treatment interruption, or having a confirmed HIV RNA ≥1,000 copies)
5. Cohort 1: suspected to have an active infection
6. Cohort 2: not suspected to have or being evaluated for an active infection

Exclusion Criteria:

1. Unlikely to attend regular clinic visits
2. History of recent talaromycosis or histoplasmosis infection currently on antifungal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients age ≥18 years with advanced HIV disease who have a CD4 count ≤100 cells/mm3 within the past 3 months, who are admitted to hospitals with a suspected infection (Cohort 1) or who are asymptomatic and registered in HIV outpatient clinic (Cohort 2) in Vietnam
Sampling Method: Non-Probability Sample
Enrollment: 1411 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of microscopy and/or culture-confirmed talaromycosis | over six to twelve months
  Cumulative incidence of microscopic and or culture-confirmed talaromycosis over six to twelve months will be recorded

SECONDARY OUTCOMES:
Incidence of other major HIV-associated opportunistic infections | over six to twelve months
  Opportunistic infections to be recorded include: tuberculosis, cryptococcosis, and histoplasmosis
Incidence of stage III and IV AIDS events | over six to twelve months
  Cumulative incidence of HIV stage III and IV event according to WHO criteria
Hospitalizations in the subsequent six to twelve months | over six to twelve months
  Cumulative incidence of hospitalizations
Mortality in the subsequent six months (Cohort 1) and twelve months (Cohort 2) | over six to twelve months
  All cause mortality will be recorded
Incidence of loss to follow up | over six to twelve months
  Loss of follow up is defined as missing >3 consecutive clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Le, MD, Principal Investigator — Duke University
Locations (2):
- Vietnam (2):
  - Hospital for Tropical Diseases, Ho Chi Minh City, Ward 1 District 5
  - National Hospital for Tropical Diseases, Hà Nội

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thu NTM, Chan JFW, Ly VT, Ngo HT, Hien HTA, Lan NPH, Chau NVV, Cai JP, Woo PCY, Day JN, van Doorn R, Thwaites G, Perfect J, Yuen K, Le T. Superiority of a Novel Mp1p Antigen Detection Enzyme Immunoassay Compared to Standard BACTEC Blood Culture in the Diagnosis of Talaromycosis. Clin Infect Dis. 2021 Jul 15;73(2):e330-e336. doi: 10.1093/cid/ciaa826. PMID 32564074